CLINICAL TRIAL: NCT04543110
Title: Neoadjuvant Immune-Modulating Radiation With Durvalumab (MEDI4736) Prior to Radical Cystectomy in Patients With Muscle-Invasive Bladder Carcinoma (RADIANT)
Brief Title: Radiation and Durvalumab Immunotherapy As Neoadjuvant Treatment for MIBC
Acronym: RADIANT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Cross Cancer Institute (Other); Hamilton Health Sciences Corporation (Other); London Health Sciences Centre (Other); Ontario Institute for Cancer Research (Other); AstraZeneca (Industry); Ozmosis Research Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OTT-19-07/OZM-105
Record Dates: First submitted 2020-07-24; First posted 2020-09-09 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Bladder Cancer
Keywords: Urothelial Carcinoma; Muscle-Invasive Bladder Cancer; Neoadjuvant; Radiation; Durvalumab; Immunotherapy
MeSH Terms: conditions — Urinary Bladder Neoplasms; Carcinoma, Transitional Cell | interventions — durvalumab

STUDY DESIGN:
Intervention Model Description: Single-arm Phase II Fleming
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Single Arm (Experimental): Immune-Modulating Radiation with Durvalumab prior to Radical Cystectomy in Patients With Muscle-Invasive Bladder Carcinoma
  Interventions: Drug: Durvalumab; Radiation: Immune Modulating Radiation

INTERVENTIONS:
Drug: Durvalumab — Durvalumab prior to Radical Cystectomy in Patients With Muscle-Invasive Bladder Carcinoma
  Other Names: (MEDI4736)
Radiation: Immune Modulating Radiation — Neoadjuvant Immune-Modulating Radiation prior to Radical Cystectomy in Patients With Muscle-Invasive Bladder Carcinoma
  Other Names: Neoadjuvant Immune Modulating Radiation

SUMMARY:
This study assesses the effect of sequential radiation and durvalumab immunotherapy given as treatment prior to surgery with radical cystectomy for bladder cancer.

DETAILED DESCRIPTION:
In this phase II study, patients who are either not eligible or declined to have chemotherapy prior to surgery for muscle-invasive bladder cancer may consent and enrol to study. Patients will have single 8 Gy hypofractionated radiation to bladder followed by 3 cycles of durvalumab immunotherapy prior to radical cystectomy. This study will assess the safety and tolerability, pathological and radiological response, and immune biological correlatives to understand the effect of radiation and durvalumab.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is willing and able to provide written informed consent
2. Patient is willing and able to comply with the protocol
3. Age ≥ 18 years
4. Body weight >30 kg.
5. Histopathologically confirmed transitional cell carcinoma/urothelial carcinoma (TCC/UC).

   1. Patients with mixed transitional/non-transitional cell histologies (adenocarcinoma, squamous cell) or variant transitional histology (eg, micropapillary, plasmacytoid, sarcomatoid, nested variant, lymphoepithelioid, nested variant) are eligible.
   2. Patients with pure non-transitional cell variant histologies and/or any component of small cell histology are not eligible.
6. Clinical stage T2-T4a N0 M0 TCC/UC, as evaluated by CT, MRI and/or PET (per standard local imaging practices) within 4 weeks prior to randomization.
7. Fit and planned for cystectomy (according to local guidelines).
8. Ineligible for neoadjuvant cisplatin-based chemotherapy OR patient declines to receive neoadjuvant cisplatin-based chemotherapy

   a) Ineligibility for chemotherapy include any of: i) Poor renal function (GFR < 50 ml/min) ii) Poor performance status (ECOG PS ≥ 2) iii) Significant (grade ≥2) neuropathy iv) Significant (grade ≥2) hearing loss v) Heart failure (NYHA-class-III/IV) OR b) Declining to receive neoadjuvant cisplatin regimen is documented by consultation with medical oncologist
9. Deemed by investigator to be medically fit (at the time of enrollment) for:

   1. Radiotherapy to pelvis
   2. Immunotherapy with durvalumab
   3. Radical cystectomy
10. Representative formalin-fixed paraffin-embedded (FFPE) tumor specimens (blocks preferred) or at least 15 unstained slides, with an associated pathology report
11. ECOG performance status of 0-1
12. Adequate hematologic and end-organ function tests.

    1. Hemoglobin ≥9.0 g/dL
    2. Absolute neutrophil count ≥1.5×109/L
    3. Platelet count ≥100×109/L
    4. Serum bilirubin ≤1.5×the upper limit of normal (ULN).

    i) This will not apply to patients with confirmed Gilbert's syndrome, who will be allowed after discussion with the study sponsor / medical monitor.

    e) Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3.0×ULN f) CrCl >40 mL/min calculated by Cockcroft-Gault equation (using actual body weight) or measured by 24-hour urine collection for determination. In cases where both are performed, measured 24- hour urine collection will be used to determine eligibility, providing an adequate collection was performed.
13. Must have a life expectancy of at least 12 weeks at enrollment
14. Patients of childbearing / reproductive potential should use highly effective birth control methods, as defined by the investigator, during the study treatment period and for a period of at least 90 days after the last dose of durvalumab. A highly effective method of birth control (as defined in Section 8.7.2) are those that result in low failure rate (i.e. less than 1% per year) when used consistently and correctly.
15. Women of child bearing potential (WOCBP) must have a negative serum (or urine) pregnancy test at the time of screening. WOCBP is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy or bilateral salpingectomy) and is not postmenopausal. Menopause is defined as 12 months of amenorrhea in a woman over age 45 years in the absence of other biological or physiological causes. In addition, females under the age of 55 years must have a serum follicle stimulating hormone, (FSH) level > 40 mIU/mL to confirm menopause.
16. Females must not be breastfeeding at time of enrollment until at least 90 days after last dose of durvalumab
17. Male patients should agree to not donate sperm during the study until at least 90 days after the last dose of durvalumab

Exclusion Criteria:

1. Evidence of suspected metastatic lymph node(s) (defined as short axis measurement of ≥10 mm as per IV contrast-enhanced CT or MRI scan) and/or PET-CT scan
2. Extravesical TCC/UC that invades the pelvic and/or abdominal wall for bladder cancer (T4b)
3. Distantly metastatic TCC/UC
4. Primary non-bladder (ie, ureter, urethral, or renal pelvis) TCC/UC
5. Inoperable tumor(s) with fixation to the pelvic wall on clinical exam
6. History of allogeneic organ transplantation that requires use of immunosuppressive agents. Patients with a history of allogenic stem cell transplantation are also excluded.
7. Malignancies other than TCC/UC within 5 years prior to Cycle 1, Day 1, with the exception of those with a negligible risk of metastasis or death and treated with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, or ductal carcinoma in situ treated surgically with curative intent) or localized prostate cancer treated with curative intent and absence of prostate-specific antigen (PSA) relapse or incidental prostate cancer (Gleason score ≤ 3 + 4 and PSA < 10 ng/mL undergoing active surveillance and treatment naive).
8. Any history of autoimmune disease or connective tissue disorder including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, glomerulonephritis, or scleroderma.

   a) The following are exceptions to this criterion: i) Patients with vitiligo or alopecia ii) Patients with hypothyroidism (eg, following Hashimoto syndrome) stable on thyroid replacement iii) Any chronic skin condition that does not require systemic therapy iv) Patients with celiac disease controlled by diet alone may be included after consultation the study sponsor and medical monitor v) Patients without active autoimmune disease in the last 5 years may be included after consultation with the study sponsor and medical monitor
9. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis testing in line with local practice), hepatitis B (known positive hepatitis B virus [HBV] surface antigen [HBsAg] result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV ribonucleic acid (RNA).
10. Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria

    a) Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after discussion with the study sponsor / medical monitor.
11. History of idiopathic pulmonary fibrosis
12. History of active primary immunodeficiency
13. Evidence of significant uncontrolled concomitant disease that could affect compliance with the protocol or interpretation of results, including significant liver disease (such as cirrhosis, uncontrolled major seizure disorder)
14. Significant cardiovascular disease, such as New York Heart Association cardiac disease (Class II or greater), myocardial infarction within 6 months prior to enrolment, unstable arrhythmias, or unstable angina.
15. Severe infections within 4 weeks prior to enrolment in the study including but not limited to hospitalization for complications of infection, bacteraemia, or severe pneumonia.
16. Major surgical procedure within 4 weeks prior to enrolment or anticipation of need for a major surgical procedure during the course of the study other than for diagnosis.
17. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
18. Known hypersensitivity or allergy to biopharmaceuticals produced in Chinese hamster ovary cells or any component of the durvalumab formulation
19. History of any illness or disease that would significant compromise patient ability to receive radiation or any reason that would preclude a patient from radiation therapy as delivered by this study design
20. Prior systemic treatment for TCC/UC

    a) Prior local intravesical chemotherapy or immunotherapy (e.g. BCG) is allowed if completed at least 6 weeks prior to initiation of study treatment
21. Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer- related conditions (eg, hormone replacement therapy) is acceptable.
22. Prior exposure to immune-mediated therapy (with exclusion of Bacillus-Calmette Guerin [BCG]), including but not limited to other anti-CTLA-4, anti-PD-1, anti-PD-L1, or anti-PD-L2 antibodies.
23. Receipt of live attenuated vaccine within 30 days prior to the first dose of IP.

    Note: Patients, if enrolled, should not receive live vaccine while receiving IP and up to 30 days after the last dose of IP.
24. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion:

    1. Intranasal, inhaled, topical steroids, or local steroid injections (eg, intra-articular injection)
    2. Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
25. Prior pelvic radiotherapy treatment
26. Treatment with any other investigational agent or participation in another clinical trial with therapeutic intent within 28 days prior to enrolment
27. Concurrent enrollment in another clinical study unless it is non- interventional or during the follow-up period of an interventional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2021-01-29 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response (pCR) Rate | Up to 2 years
  pCR rate is defined as the proportion of patients whose pathological staging was T0N0M0 as assessed using specimens obtained post radical cystectomy following the study intervention.

SECONDARY OUTCOMES:
Adverse events | Up to 2 years
  Adverse events related to the study treatment will be identified and characterized using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. A copy of the CTCAE version 5.0 can be downloaded from the Cancer Therapy Evaluation Program website (http://ctep.cancer.gov). Data will be collected from time of confirmed study entry
Rate of delay of surgery | Up to 2 years
  Feasibility. Surgery is expected to occur within 90 days of radiotherapy. Any delay beyond that will be noted and the cause of the delay attributed to study intervention or otherwise, with supporting details.
Rate of Pathological Downstaging | Up to 2 years
  Proportion of patients who have pathological staging <T2 as determined after radical cystectomy.
Recurrence rates at 1 year and 2 years | Up to 2 years
  he proportion of patients who have radiographically confirmed recurrence of their cancer at 1 and 2 years. Time to recurrence is defined from the time of study entry to the first recurrence of disease after cystectomy. A recurrence of disease includes local (pelvic) recurrence, urinary tract recurrence, or distant metastases of urothelial carcinoma. Recurrence rate will be assessed using computed tomography (CT)/magnetic resonance imaging (MRI) and/or Positron Emission Tomography (PET)-CT (per standard local imaging practices) and pathology testing performed according to local standards and as clinically indicated.
Overall survival rate at 1 and 2 years | Up to 2 years
  The proportion of patients who are alive at 1 and 2 years. Overall survival is defined from the date of study entry until death of any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Ong, MD, Principal Investigator — Ottawa Hospital Research Institute; Naveen Basappa, MD, Principal Investigator — Cross Cancer Institute
Locations (4):
- Canada (4):
  - Cross Cancer Institute, Edmonton, Alberta
  - Juravinski Cancer Centre, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: No
Qualified researchers can contact Dr. Michael Ong regarding sharing of data and be evaluated for what their purpose and plan is for the data.